CLINICAL TRIAL: NCT01103700
Title: Evaluation of Multidisciplinary Palliative Care on Terminal Cancer Patients in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Shao-Yi Cheng/Attending Physician, Department of Family Medicine
Other Study IDs: 201003030R
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2010-04

CONDITIONS: Cancer
Keywords: Quality of dying and death of terminal cancer patients
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study is to compare the quality of dying and death of terminal cancer patients from the perspectives of medical staff and main care giver (family). The hypothesis is that their view points will be different.

ELIGIBILITY:
Inclusion Criteria:

* Cognitively intact.
* Contact with the patient in the last month.

Exclusion Criteria:

* Cognitively not intact.
* No contact with the patient in the last month.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Main care givers of deceased patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-07 (Estimated); Study Completion 2010-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Yi Cheng, MD, MSc, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan, Taiwan